CLINICAL TRIAL: NCT05921916
Title: Randomized, Double Blind, Placebo Controlled "First-in-human" Study to Assess the Safety and Tolerability of Single Ascending Oral Doses and Multiple Oral Doses of MBF-118 in Healthy Young Volunteers
Brief Title: Study to Assess the Safety and Tolerability of MBF-118 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medibiofarma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MBF-118CT-01; 2019-002967-80 (EudraCT Number)
Record Dates: First submitted 2023-06-14; First posted 2023-06-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: PPAR gamma partial agonist; anti-inflammatory; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single center, randomized, double-blind, placebo-controlled clinical study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- MBF-118 100mg oral single dose (Experimental): Drug: MBF-118 100mg oral capsules single dose Hard gelatin capsules
  Interventions: Drug: MBF-118 oral capsules
- MBF-118 200 mg oral single dose (Experimental): Drug: MBF-118 200mg oral capsules single dose Hard gelatin capsules
  Interventions: Drug: MBF-118 oral capsules
- MBF-118 400 mg oral single dose (Experimental): Drug: MBF-118 400mg oral capsules single dose Hard gelatin capsules
  Interventions: Drug: MBF-118 oral capsules
- MBF-118 100 mg oral multiple dose (Experimental): Drug: MBF-118 100mg oral capsules multiple dose. One single daily dose during five days.
  Hard gelatin capsules
  Interventions: Drug: MBF-118 oral capsules
- MBF-118 200 mg oral multiple dose (Experimental): Drug: MBF-118 200mg oral capsules multiple dose. One single daily dose during five days.
  Hard gelatin capsules
  Interventions: Drug: MBF-118 oral capsules
- MBF-118 400 mg oral multiple dose (Experimental): Drug: MBF-118 400mg oral capsules multiple dose. One single daily dose during five days.
  Hard gelatin capsules
  Interventions: Drug: MBF-118 oral capsules
- Placebo oral single dose (Placebo Comparator): Placebo: Hard gelatin capsules single dose
  Interventions: Drug: Placebo oral capsule
- Placebo oral multiple dose (Placebo Comparator): Placebo: Hard gelatin capsules. One single daily dose during five days.
  Interventions: Drug: Placebo oral capsule
- MBF-118 600 mg oral single dose (Experimental): Drug: MBF-118 600mg oral capsules single dose Hard gelatin capsules
  Interventions: Drug: MBF-118 oral capsules

INTERVENTIONS:
Drug: MBF-118 oral capsules — MBF-118 oral capsules PPAR gamma receptor partial agonist
  Arms: MBF-118 100 mg oral multiple dose; MBF-118 100mg oral single dose; MBF-118 200 mg oral multiple dose; MBF-118 200 mg oral single dose; MBF-118 400 mg oral multiple dose; MBF-118 400 mg oral single dose; MBF-118 600 mg oral single dose
Drug: Placebo oral capsule — Placebo oral capsule solid microcrystalline cellulose
  Arms: Placebo oral multiple dose; Placebo oral single dose

SUMMARY:
This is a single center, randomised, double blind, placebo controlled clinical study to assess the safety and tolerability of MBF-118 in healthy volunteers.This clinical phase I trial is divided in two stages and involves, first, a single ascending dose (SAD) study in healthy young male volunteers and then a multiple ascending dose (MAD) study in healthy young men and woman. MBF-118 is developed for the treatment of cancer.

DETAILED DESCRIPTION:
This clinical phase I trial is divided in two stages. The first stage will be a dose escalation study without therapeutic benefit, in which MBF-118 will be administered as single oral ascending dose to healthy young male volunteers. Up to four different rising doses will be tested (100 mg, 200 mg, 400 mg and 600 mg) in groups/cohorts of 8 participants. Thus, four groups/cohorts will participate. For each dose level/group, the participants will be randomized to active or placebo with 2 participants being randomly assigned to placebo and 6 to the active drug. First, one volunteer will receive active drug (subgroup 1); after at least 72h of safety and tolerability assessment a second subgroup of 3 volunteers will receive 2 active drug and 1 placebo; after at least another 72h of safety and tolerability parameters assessment a third subgroup of 4 volunteers will receive 3 active drug and 1 placebo. After evaluation of safety parameters of corresponding dose level, the process will replicate one week afterwards in the following dosages.

The second stage will be a dose escalation study without therapeutic benefit, in which MBF-118 will be administered as single oral daily dose, during 5 days to young male and female healthy volunteers. Up to three different rising dose levels will be tested (100 mg, 200 mg, and 400 mg) in cohorts of 8 subjects that are randomised to active treatment and placebo (6:2) and divided into three subsequent treatment blocks, as described above in the first stage.

The pharmacokinetics profile of MBF-118 will be also assessed at each dose level tested of the Single ascending dose study and the multiple ascending dose study.

ELIGIBILITY:
Inclusion Criteria:

To be included in the single dose study, subjects should meet all the following criteria at the screening visit:

1. Healthy male subjects, 18-45 years (inclusive) of age at the time of enrolment.
2. Body weight within normal range (Quetelet's index between 19 and 27) expressed as weight (kg) / height (m2).
3. Normal clinical records and physical examination.
4. Laboratory tests (hematology and biochemistry) within the range of normal values, according to the Biochemistry laboratory reference values of the 'Hospital de la Santa Creu i Sant Pau'. Variations may be admitted according to the clinical criteria of the CIM-Sant Pau.
5. Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ DBP between 50-90 mm Hg / HR between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
6. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner using some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
7. To be able to understand the nature of the study and comply with all their requirements.
8. Free acceptance to participate in the study should be stated in an informed consent document signed by the volunteer which must be approved by the CREC.

For the multiple dose study in healthy male and female volunteers, subjects meeting all the following inclusion criteria at screening visit:

1. Healthy male and female subjects, 18-45 years (inclusive) of age at the time of enrolment.
2. Body weight within normal range (Quetelet's index between 19 and 27) expressed as weight (kg) / height (m2).
3. Normal clinical records and physical examination at screening and baseline.
4. Laboratory tests (hematology, biochemistry and urianalysis) within the range of normal values, according to the laboratory reference values of the 'Hospital de la Santa Creu i Sant Pau'. Variations may be admitted according to the clinical criteria of the CIM-Sant Pau.
5. Clinically acceptable temperature, blood pressure and pulse rate in supine and standing position (SBP between 100-140 mm Hg/ DBP between 50-90 mm Hg / HR between 50-100 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
6. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner using some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
7. To be able to understand the nature of the study and comply with all their requirements.
8. Free acceptance to participate in the study by obtains signed informed consent form approved by the CREC.
9. Females must be of non childbearing potential (i.e. surgically sterile) or have to use contraceptive measures ( non-hormonal) such as condom, diaphragm or cervical / vault caps with spermicide until 28 days post administration

Exclusion Criteria:

* For the single dose study and multiple dose study meeting any of the following criteria at screening visit will be excluded from entry into the study:

  1. History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 g/day for men and >24g/day for women
  2. Heavy consumer of stimulating beverages (>5 coffees, teas, chocolate or cola drinks per day) and grape juice.
  3. Background of idiosyncrasy, food intolerance, hypersensitivity or adverse reactions to any drug or Galenical form.
  4. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
  5. Intake of any medication within 2 weeks prior taking the study treatment (except for use of paracetamol in short-term symptomatic treatments), including over-the-counter products (including natural food supplements, vitamins and medicinal plants products), or any enzymatic inductor or inhibitor within 3 months before the drug administration.
  6. Positive serology for hepatitis B, C or HIV.
  7. Background or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological disease or other chronic diseases.
  8. History of psychiatric diseases or epileptic seizures.
  9. 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
  10. Having undergone major surgery during the previous 6 months.
  11. Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc.) from 6 months prior to drug administration.
  12. Participation in other clinical trials during the previous 90 days (drug to drug period) in which an investigational drug or a commercially available drug was tested.
  13. Donation of blood during the 4 weeks preceding the drug administration.
  14. Severe or moderate acute illness 4 weeks before drug administration.
  15. Clinically significant abnormal laboratory values (as determined by the PI) at the screening evaluation.
  16. Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract
  17. Positive results of the drugs at screening period or the day before starting treatment period. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the PI).
  18. Female with positive results from pregnancy test or breast-feeding ( only in MAD stage)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | Day 1 through Day 5
  Classification based in the Medical Dictionary for Regulatory Activities (MedDRa) Adverse Events will be qualified according to the definitions and values stated in CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Joan Martinez, MD, Principal Investigator — CIM-Sant Pau Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- CIM-Sant Pau Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Spain